CLINICAL TRIAL: NCT01891942
Title: Influence of Trigger Threshold on Controlled Twitch Mouth Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, DM Hua, Influence of Trigger Threshold on Controlled Twitch Mouth Pressure, Guangzhou Institute of Respiratory Disease
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Diagnostic
Other Study IDs: GIRD-566; GIRD-566 (Registry Identifier: GuangzhouIRD)
Record Dates: First submitted 2013-06-26; First posted 2013-07-03 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-06

CONDITIONS: COPD; Healthy
Keywords: Normal; subjects
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- COPD patients (Experimental): All of the COPD patients included in this study were stable with no episodes of exacerbation within the previous 2 months. Patients with COPD were not currently being treated with oral corticosteroids.
  Interventions: Procedure: twitch by magstim
- normal subjects (Experimental): Fifteen healthy men with normal lung function
  Interventions: Procedure: twitch by magstim

INTERVENTIONS:
Procedure: twitch by magstim

SUMMARY:
The inspiratory pressure trigger is essential when assessing the twitch mouth pressure (Tw Pmo) for avoiding glottic closure. However, the difference in inspiratory pressure trigger threshold may influence the values of Tw Pmo. We sought to determine the trigger threshold for healthy subjects and COPD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of COPD
2. Stable with no episodes of exacerbation within the previous 2 months
3. Do not currently being treated with oral corticosteroids

Exclusion Criteria:

1. Not stable within the previous 2 months.
2. Patients with COPD were currently being treated with oral corticosteroids

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Twitch mouth pressure | 2 weeks

SECONDARY OUTCOMES:
Twitch oesophageal pressure | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rong-chang Chen, Master, Study Chair — Guangzhou Instiute of Respiratory Disease; Dong-ming Hua, Master, Principal Investigator — Guangzhou Institue of Respiratory Disease; Nan-shan Zhong, Bachelor, Study Chair — Guangzhou Institue of Respiratory Disease
Locations (1):
- Guangzhou Institute Respiratory Disease, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Walker DJ, Ertl T, Walterspacher S, Schlager D, Roecker K, Windisch W, Kabitz HJ. Respiratory muscle function during a six-week period of normocapnic hyperpnoea training. Respir Physiol Neurobiol. 2013 Aug 15;188(2):208-13. doi: 10.1016/j.resp.2013.05.005. Epub 2013 May 17. PMID 23689008
- [Result] Hua DM, Liang YH, Xie YK, Liu Q, Zheng ZG, Chen RC, Zhong NS. Use of twitch mouth pressure to assess diaphragm strength in patients with chronic obstructive pulmonary disease. Respir Physiol Neurobiol. 2013 Jul 1;187(3):211-6. doi: 10.1016/j.resp.2013.04.012. Epub 2013 Apr 15. PMID 23597835